CLINICAL TRIAL: NCT05631678
Title: An Open-lable, Two- Period, Single-sequence, Self-controlled Study to Evaluate the Effect of Oral Rifampicin or Itraconazole on the Pharmacokinetics of ASK120067 Tablets
Brief Title: Drug-drug Interaction Study Beteewn ASK120067 and Rifampicin or Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASK120067-PK-1
Record Dates: First submitted 2022-11-11; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the effect of oral rifampicin on the pharmacokinetics of ASK120067 tablets (Experimental): Take ASK120067 tablets orally once on the first day at 160mg in fast condition；Take rifampicin capsules orally once on the days 8 to 17 at 600mg in fast condition, and a combination of 160mg ASK120067 and 600mg rifampicin were administrated on the 15th day in fast condition.
  Interventions: Drug: Rifampicin; ASK120067
- effect of oral itraconazole on the pharmacokinetics of ASK120067 tablets (Experimental): Take ASK120067 tablets orally once on the first day at 80mg in fast condition；Take itraconazole capsules orally twice on the days 8 to 13 at 200mg in fed condition, and a combination of 80mg ASK120067 and 200mg itraconazole were administrated on the 11th day in fast condition.
  Interventions: Drug: ASK120067;itraconazole

INTERVENTIONS:
Drug: Rifampicin; ASK120067 — Take ASK120067 tablets orally once on the first day at 160mg in fast condition;Take rifampicin capsules orally once on the days 8 to 17 at 600mg in fast condition, and a combination of 160mg ASk120067 and 600mg rifampicin were administrated on the 15th day in fast condition.
  Arms: the effect of oral rifampicin on the pharmacokinetics of ASK120067 tablets
Drug: ASK120067;itraconazole — Take ASK120067 tablets orally once on the first day at 80mg in fast condition;Take itraconazole capsules orally twice on the days 8 to 13 at 200mg in fed condition, and a combination of 80mg ASK120067 and 200mg itraconazole were administrated on the 11th day in fast condition.
  Arms: effect of oral itraconazole on the pharmacokinetics of ASK120067 tablets

SUMMARY:
To evaluate the effects of oral administration rifampicin or itraconazole capsules on the pharmacokinetics of ASK120067 and its metabolite CCB4580030 in healthy subjects.

To evaluate the safety of ASK120067 tablets or combination with rifampicin capsules or itraconazole capsules in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult subjects, male and female;
2. Age: 18-45 years old (including boundary value);
3. Body weight: body mass index (BMI) between 18.5 and 26.0 kg/m2 (including boundary values);
4. Subjects are willing to sign the informed consent;
5. Subjects are able to communicate well with investigators and complete the clinical trial in according to the protocol.

Exclusion Criteria:

1. patients with clinical significance who are abnormal by comprehensive physical examination, vital signs examination, routine laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function), 12-lead electrocardiogram, and positive and lateral chest radiographs;
2. HBSAg HCVAb HIVAb, and treponema palliatum antibody test results were positive;
3. taking any drugs that inhibit or induce hepatic metabolism of drugs (especially CYP3A4, CYP2C8, CYP2C9 and CYP2C19) within 30 days before the screening period (e.g., inducers - barbiturates, carbamazepine, phenytoin, rifampicin, glucocorticoids, rifabutin, PPI inhibitors; Inhibitors: SSRI antidepressants, cimetidine, diltiazem, macrolides, verapamil, nitroimidazoles, sedative hypnotics, fluoroquinolones, antihistamines);'
4. taking any medication 14 days before the trial;
5. taking any investigational drug or participating in any investigational drug within 3 months before the screening period;
6. previous history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torssion ventricular tachycardia, ventricular tachycardia, long QT syndrome or symptoms of long QT syndrome and family history (genetic proof or sudden death of a close relative at young age);
7. major surgery within 6 months before the screening period or surgical incision did not heal completely;
8. history of any clinically serious illness or disease or condition considered by the investigators to be likely to affect the results of the trial, including but not limited to a history of cardiac, respiratory, endocrine, nervous, digestive, urinary, or hematologic, immunologic, psychiatric, or metabolic diseases;
9. specific allergic history (asthma, measles, eczema, etc.) or allergic constitution (presence of two or more allergens), or allergic to EGFR receptor inhibitor drugs or any component of the trial drugs; allergic to any food ingredients or have special requirements for diet and cannot abide by the uniform diet;
10. smoking more than 5 cigarettes per day within 3 months before screening period and unable to quit during the trial;
11. Heavy drinking or regular drinking within 3 months before the screening period, defined as drinking more than 14 units of alcohol per week (1 unit =360ml of beer or 45 ml of 40% spirits or 150 ml of wine); Or alcohol breath test > 0.0mg /100mLduring screening;
12. history of drugs use or drugs abuse screening positive;
13. special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or drank excessive tea, coffee, grapefruit/grapefruit juice and/or caffeinated beverages (more than 8 cups per day, 200 mL per cup on average) within 2 weeks before the first dose of research medication;
14. Pregnant or lactating women, or pregnancy screening positive;
15. Sujects plan to have a child during the trial or within 6 months after completion of the trial, or do not agree that heself /herself and his/her spouse use strict contraception (condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, or other contraceptive methods) during the trial and within 6 months after completion of the trial.
16. History of lost blood or donated a blood volume of 400 mL within 3 months before the screening period or planing to donate blood within 1 month after the end of the trial;
17. Subjects were vaccinated within 15 days before screening or planing to be vaccinated during the trial, or have not been vaccinated against COVID-19;
18. Subjects may be unable to complete the study for other reasons or may be considered inappropriate by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out maximum concentration
AUC | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Tmax | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out time to reach maximum concentration
t1/2 | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Blood samples will be collected from each subject at pre-specified times after the administration of ASK120067 in each period, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
CL/F | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out apparent clearance
Vd/F | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out apparent volume of distribution
λz | Blood samples will be collected from each subject after the administration of ASK120067 on Day 1 and Day 15 in arm A ,and on Day 1 and Day 11 in arm B (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 h post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points after the administration of ASK120067 in each period to figure out apparent terminal elimination rate constant
Incidence and Severity of Treatment-Emergent Adverse Events | Adverse events will be collected from baseline until 18 days of arm A or 14 days of arm B after the first dose administration and the follow-up period
  Assessed by number and severity of adverse events as recorded on the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Principal Investigator — Drum Tower Hospital of Nanjing University School of Medical
Locations (1):
- Drum Tower Hospital of Nanjing University School of Medical, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cao B, Huang L, Liu M, Lin H, Ma T, Zhao Y, Geng Y, Yang Y, Guo H, Li J. Phase 1 study to evaluate the effects of rifampin or itraconazole on the pharmacokinetics of limertinib (ASK120067), a novel mutant-selective inhibitor of the epidermal growth factor receptor in healthy Chinese subjects. Expert Opin Drug Metab Toxicol. 2023 Sep;19(9):653-664. doi: 10.1080/17425255.2023.2260738. Epub 2023 Oct 12. PMID 37811634